CLINICAL TRIAL: NCT00737542
Title: A Prospective Randomized Double-blind, Placebo-controlled Study of the Effect of Preoperative Analgesia With Local Lidocaine Infiltration for Pain Management Post Cesarean Delivery.
Brief Title: Local Lidocaine Infiltration for Pain Management Post Cesarean Delivery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Roy Kessous Md., Soroka University Medical Center
Other Study IDs: sor470408CTIL
Record Dates: First submitted 2008-08-17; First posted 2008-08-19 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2008-08

CONDITIONS: Pain; Cesarean Delivery
Keywords: management; post
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Chloride

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: NACL 0.9%
- B (Experimental)
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine
  Arms: B
Drug: NACL 0.9%
  Arms: A

SUMMARY:
The objective of this prospective, double-blinded, placebo-controlled, randomized study is to evaluate the impact of preemptive analgesia using incisional site infiltration of lidocaine as compared to saline solution on post operative pain control in women undergoing cesarean deliveries.

DETAILED DESCRIPTION:
The studied population would be based on women who are scheduled for an elective cesarean delivery under general/spinal analgesia using a transverse lower abdominal incision.

Prior to each operation, the surgeon will be provided with a syringe containing a 20 mL solution of 1% lidocaine or 0.9% sodium chloride, which will be injected subcutaneously to the incisional site region after anesthesia and before the beginning of the surgery.

After the operation the conventional post cesarean analgesic regime will be used and recorded for all women.

The self-report of pain will be assessed by the patient using a validated visual analog scale, as instructed by the nursing staff.

The patient's mark will be used as a numerical index of pain intensity. The reports will be taken by the patients in intervals of 4 hours for 48 hours after the operation. In addition, analgesic requirements of the patient will be monitored and recorded by the nursing staff and used for comparison between the two study group

ELIGIBILITY:
Inclusion Criteria:

* Women who are scheduled for an elective cesarean delivery under general/spinal analgesia using a transverse lower abdominal incision.

Exclusion Criteria:

* More than two previous cesarean deliveries
* Other abdominal operations in the past
* Morbid obesity
* Diabetes mellitus, neurological diseases, systemic vascular disease.
* Mental disability
* Lidocaine sensitivity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Obstetrics and Gynecology - Soroka University Medical Center, Beersheba, Israel